CLINICAL TRIAL: NCT04657497
Title: A Placebo-controlled, Multicenter, Double-blind, Randomized, Parallel-group Comparative Study in SARS-CoV-2 Infection (COVID-19)
Brief Title: A Study of FOY-305 in Patients With SARS-Cov-2 Infection (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOY-305-01
Record Dates: First submitted 2020-11-09; First posted 2020-12-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV-2 Infection (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOY-305 group (Experimental): Camostat Mesilate tablets 600 mg will be orally administered 4 times daily, before breakfast, before lunch, before evening meal, and at bedtime. The treatment period is up to 14 days.
  Interventions: Drug: FOY-305
- Placebo group (Placebo Comparator): Placebo tablets will be orally administered 4 times daily, before breakfast, before lunch, before evening meal, and at bedtime. The treatment period is up to 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FOY-305 — Specified Dosage and Duration of Treatment
  Arms: FOY-305 group
Drug: Placebo — Specified Dosage and Duration of Treatment
  Arms: Placebo group

SUMMARY:
To assess the efficacy and safety of FOY-305 in patients with SARS-CoV-2 infection (COVID-19) in a placebo-controlled, multicenter, double-blind, randomized, parallel-group comparative study.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient or outpatient: Inpatient
2. Positive SARS-CoV-2 test by a method eligible for definitive diagnosis
3. Enrollment in this study within 5 days after onset of symptoms of SARS-CoV-2 infection (COVID-19) (for asymptomatic patients, enrollment in this study within 5 days after collection of the sample that tested positive)

Exclusion Criteria:

1. Receiving oxygen therapy
2. Difficulty in swallowing oral medication
3. History of COVID-19
4. History of vaccination against COVID-19
5. Taking camostat mesilate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Time to SARS-CoV-2 negative test | Up to 14 days
  Time to SARS-CoV-2 negative test as assessed by the local laboratory

SECONDARY OUTCOMES:
Time to SARS-CoV-2 negative test | Up to 14 days
  Time to SARS-CoV-2 negative test as assessed by the central laboratory
Proportion of subjects who test negative for SARS-CoV-2 | Up to 14 days
  Proportion of subjects who test negative for SARS-CoV-2 (as assessed by the local and central laboratories)
Ordinal scale for severity | Up to 14 days
  Ordinal scale for severity. The minimum score is 0: No clinical or virological evidence of infection, representing the better outcome, and the maximum value is 8: Death, representing the worse outcome.
Proportion of subjects on mechanical ventilator | Up to 14 days
  Proportion of subjects on mechanical ventilator
Survival status (alive/death) | Up to 14 days
  Proportion of subjects alive or death

CONTACTS AND LOCATIONS:
Overall Officials: Naoyuki Komura, Study Director — Ono Pharmaceutical Co. Ltd
Locations (25):
- Japan (25):
  - Aichi Clinical Site 1, Tokoname, Aichi-ken
  - Chiba Clinical Site 1, Narita, Chiba
  - Fukuoka Clinical Site 1, Ōkawa, Fukuoka
  - Ibaraki Clinical Site 1, Tsuchiura, Ibaraki
  - Ishikawa Clinical Site 1, Kanazawa, Ishikawa-ken
  - Kanagawa Clinical Site 3, Kawasaki, Kanagawa
  - Kanagawa Clinical Site 1, Yokohama, Kanagawa
  - Kanagawa Clinical Site 2, Yokosuka, Kanagawa
  - Mie Clinical Site 1, Yokkaichi, Mie-ken
  - Niigata Clinical Site 1, Nagaoka, Niigata
  - Osaka Clinical Site 2, Daitō, Osaka
  - Saitama Clinical Site 3, Kawagoe, Saitama
  - Saitama Clinical Site 1, Kukichūō, Saitama
  - Saitama Clinical Site 2, Kumagaya, Saitama
  - Tokyo Clinical Site 5, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site 9, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site1, Hachiōji, Tokyo
  - Tokyo Clinical Site 7, Itabashi-ku, Tokyo
  - Tokyo Clinical Site 3, Meguro-ku, Tokyo
  - Tokyo Clinical Site 4, Shinagawa-ku, Tokyo
  - Tokyo Clinical Site 8, Sibuya-ku, Tokyo
  - Tokyo Clinical Site2, Sibuya-ku, Tokyo
  - Tokyo Clinical Site 6, Tachikawa, Tokyo
  - Okayama Clinical Site 1, Okayama
  - Osaka Clinical Site 1, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinoshita T, Shinoda M, Nishizaki Y, Shiraki K, Hirai Y, Kichikawa Y, Tsushima K, Shinkai M, Komura N, Yoshida K, Kido Y, Kakeya H, Uemura N, Kadota J. A multicenter, double-blind, randomized, parallel-group, placebo-controlled study to evaluate the efficacy and safety of camostat mesilate in patients with COVID-19 (CANDLE study). BMC Med. 2022 Sep 27;20(1):342. doi: 10.1186/s12916-022-02518-7. PMID 36163020